CLINICAL TRIAL: NCT02984735
Title: Association Between Chewing Performance Level and Gross Motor Function in Children With Cerebral Palsy
Brief Title: Chewing Performance Level and Gross Motor Function in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Selen Serel Arslan, Hacettepe University
Other Study IDs: HACETTEPEUNI
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy; Chewing Problem; Gross Motor Development Delay
Keywords: chewing; cerebral palsy; chewing disorders; gross motor function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Evaluation of children with spastic CP: Children with a diagnosis of spastic CP aged 2 to 12 years who were referred due to chewing/swallowing problems by pediatric neurologists were included. The inclusion criteria were above the age of 24 months, and had complaints about chewing function. Children under the age of 24 months, requiring tube feeding or taking any oral nutritional supplements, and used any medicine and/or oral appliances that could affect the chewing performance, were excluded.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Descriptive characteristics including age, height and weight were recorded. Chewing performance level was determined with the Karaduman Chewing Performance Scale (KCPS). Each child was placed in a sitting position (either on a chair or on his/her mother's arm) with the head upright and with the midline position and arms and legs supported, and required to bite and chew a standardized biscuit, and no clue was given on how to chew. The physical therapist rated the chewing performance according to the KCPS. All children underwent a physical examination by a physical therapist to determine gross motor function by applying the Gross Motor Function Classification System (GMFCS). In addition to GMFCS, number of affected limbs of the children was also noted.

SUMMARY:
The purpose of this study is to determine the association between gross motor function and chewing performance level in children with cerebral palsy (CP). A cross-sectional study was conducted in 152 children (ages 2-10y, 51.3% male) with a diagnosis of spastic CP. The Gross Motor Function Classification System (GMFCS) was used to determine gross motor function levels of children. Chewing performance level was determined by using the Karaduman Chewing Performance Scale (KCPS).

DETAILED DESCRIPTION:
The purpose of this study is to determine the association between gross motor function and chewing performance level in children with cerebral palsy (CP). A cross-sectional study was conducted in 152 children (ages 2-10y, 51.3% male) with a diagnosis of spastic CP. The Gross Motor Function Classification System (GMFCS) was used to determine gross motor function levels of children. Chewing performance level was determined by using the Karaduman Chewing Performance Scale (KCPS).Children with a diagnosis of spastic CP aged 2 to 12 years who were referred due to chewing/swallowing problems by pediatric neurologists were included. The inclusion criteria were above the age of 24 months, and had complaints about chewing function. Children under the age of 24 months, requiring tube feeding or taking any oral nutritional supplements, and used any medicine and/or oral appliances that could affect the chewing performance, were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 24 months
* Having complaints about chewing function.

Exclusion Criteria:

* Under the age of 24 months
* Requiring tube feeding or taking any oral nutritional supplements
* Using any medicine and/or oral appliances

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with a diagnosis of spastic CP aged 2 to 12 years who were referred due to chewing/swallowing problems by pediatric neurologists
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Chewing performance level | 10 minutes
  Chewing evaluation

SECONDARY OUTCOMES:
Gross motor function level | 10 minutes
  Motor function evaluation

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No